CLINICAL TRIAL: NCT05205720
Title: Application of Celiac Plexus Block in Postoperative Analgesia of Whipple Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0594
Record Dates: First submitted 2021-12-29; First posted 2022-01-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative; Nerve Block
Keywords: celiac plexus block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NB group (Experimental): Celiac plexus block (CPB) was added to the postoperative analgesia plan.
  CPB: the target nerve is located in the retroperitoneal space, embedded in the fat in front of the aorta, and distributed in a network along the anterolateral wall of the aorta, just at the beginning of the celiac trunk. During direct vision (anterior) block, first expose the upper edge of the pancreas, palpate the abdominal aorta and abdominal trunk, and palpate the pulsation of the common hepatic artery and splenic artery at the level of the abdominal trunk. Use a 25g 6cm puncture needle with an extension tube and a syringe pumped back by an assistant to form a negative pressure, then the needle is inserted into the fat on both sides of the abdominal aorta. If there is no blood or fluid outflow, slowly inject 10ml of 0.5% ropivacaine each side. After pulling out the needle, observe whether there is damage and bleeding. If necessary, use low-energy electrocoagulation to stop bleeding.
  Interventions: Procedure: Celiac plexus block; Drug: Ropivacaine
- GC group (No Intervention): The same analgesic plan as the experimental group, except that CPB is not performed.

INTERVENTIONS:
Procedure: Celiac plexus block — The surgeon is instructed to perform a single celiac plexus block under direct vision. 10ml 0.5% ropivacaine is injected into the nerve in both sides.
  Arms: NB group
Drug: Ropivacaine — Mixed solution for nerve block, made of 0.75% ropivacaine (Naropin, Astrazeneca AB) diluted in different proportions.
  Arms: NB group

SUMMARY:
This subject intends to explore the value of intraoperative celiac plexus block in postoperative acute pain management and its promoting effect on patients' rapid recovery during Whipple surgery through a randomized controlled trial.

DETAILED DESCRIPTION:
This study is a single center, randomized, single-blind controlled study. After calculating the sample size, 66 subjects would be randomly assigned to nerve block group (NB group: local anesthetic injection at the target position) and blank control group (GC group: no celiac plexus block) according to the ratio of 1:1, in order to evaluate the effectiveness and safety of celiac plexus block (CPB) as a part of multimodal analgesia for postoperative pain management.

Anesthesia protocol: the standard anesthesia protocol for open Whipple surgery in our hospital was adopted.

Postoperative analgesia plan: before abdominal closure at the end of operation, The surgeon was instructed to perform a single celiac plexus block (CPB) under direct vision. Ropivacaine was injected into the target nerve in NB group, but no injection in GC group. After the operation, the anesthesiologist used ropivacaine to perform ultrasound-guided abdominal wall nerve block. When leaving the operating room, connect intravenous analgesia pump. Patients with subjective pain score of 3 or above can press. If the analgesia is insufficient, intravenous injection of dezocine can be added temporarily. The intravenous analgesia pump shall be withdrawn after 72 hours of use. If the analgesia pump is used up and is still needed, the anesthesiologist can evaluate and add medicine.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18years;
2. received open Whipple surgery.

Exclusion Criteria:

1. patients unable to cooperate with evaluations;
2. patients with history of drug abuse, local anesthetic allergy, anatomical variation of the celiac ganglia indicated by abdominal CT, abdominal aortic diseases;
3. non-standard surgical procedures, planned postoperative ICU admission;
4. American Society of Anesthesiologists (ASA) classification of 4 or 5.

Withdrawal criteria:

Patients who underwent unplanned surgeries, required reintubation or a second surgery, received ICU care within three days post-surgery, died within two weeks post-surgery, or experienced any unexpected events were withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours after surgery
  Morphine equivalent

SECONDARY OUTCOMES:
Press of the analgesic pump | Every 24 hours post-surgery for 72 hours
  Daily frequency of pump presses
Time to first flatus | 72 hours after surgery
Length of postoperative hospitalization | After surgery to before discharge, up to 2 months
White blood cell count | At the end of surgery and 24 hours post-surgery
  Laboratory tests of white blood cell count (WBC)
C-reactive protein | At the end of surgery and 24 hours post-surgery
  Laboratory tests of C-reactive protein (CRP)
Erythrocyte sedimentation rate | At the end of surgery and 24 hours post-surgery
  Laboratory tests of erythrocyte sedimentation rate (ESR)
Interleukin-6 | At the end of surgery and 24 hours post-surgery
  Laboratory tests of interleukin-6 (IL-6)
Procalcitonin | At the end of surgery and 24 hours post-surgery
  Laboratory tests of procalcitonin (PCT)
Pain scores | 6, 12, 24, 48, 72 hours after surgery
  VAS (0 indicates no pain and score 10 indicates the most severe pain)
Cardiac index changes during celiac plexus block | Before and 5、10、20 minutes after CPB
  Celiac plexus block (CPB)
Systemic vascular resistance index changes during celiac plexus block | Before and 5、10、20 minutes after CPB
  Celiac plexus block (CPB)
Postoperative mean arterial pressure | Every 12 hours post-surgery for 72 hours
  Mean arterial pressure (MAP)
Postoperative heart rate | Every 12 hours post-surgery for 72 hours
  Heart rate (HR)

CONTACTS AND LOCATIONS:
Overall Officials: Minpu Li, Master, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers whose proposed use of the data has been approved.
Supporting Information: SAP
Time Frame: With publication

REFERENCES:
- [Derived] Li M, Fang L, Xing T, Wang C, Chen S, Yu S, Zhu J. A single-blind randomized controlled trial of celiac plexus block for analgesia after whipple surgery. BMC Anesthesiol. 2025 Apr 22;25(1):193. doi: 10.1186/s12871-025-03045-7. PMID 40263988